CLINICAL TRIAL: NCT04559685
Title: A Phase 0, First in Human, Open-label Study of Intravenous Aminolevulinic Acid HCl (ALA) and MR-Guided Focused Ultrasound Device (MRgFUS) in Participants with Recurrent High Grade Glioma (HGG)
Brief Title: Study of Sonodynamic Therapy in Participants with Recurrent High-Grade Glioma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nader Sanai (Other)
Collaborators: Barrow Neurological Institute (Other); Ivy Brain Tumor Center (Other); SonALAsense, Inc. (Industry); InSightec (Industry)
Responsible Party: Sponsor-Investigator, Nader Sanai, Deputy Director, Ivy Brain Tumor Center, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11; 21-500-032-34-38 (Other: St. Joseph's Hospital and Medical Center)
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (5):
- Arm A Energy Dose-escalation (Experimental): In Arm A, the dose-escalation cohort, there will be 3 cohorts of ascending MRgFUS power/energy dose combinations with a fixed SONALA-001 dose and fixed surgical time. Arm A will determine the power/energy dose combination for Arm B.
  Interventions: Combination Product: SONALA-001(ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Arm B Time-escalation (Experimental): In Arm B, the time-escalation cohort, the SONALA-001 and power/energy dose combination will be fixed. Participants will be enrolled into two time cohorts (2 days and 6 days post-SDT).
  Interventions: Combination Product: SONALA-001(ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Arm C ALA Dose-escalation (Experimental): In Arm C, the MRgFUS power/energy dose will be fixed based on Arm A MTD/OBD, with the SONALA-001 dose escalation.
  Interventions: Combination Product: SONALA-001(ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Arm D MRgFUS alone (Experimental): In Arm D, MRgFUS treatment alone will be given at the optimal energy determined from previous Arms.
  Interventions: Device: MR-Guided Focused Ultrasound device (MRgFUS)
- Arm E Optimal energy and ALA dose (Experimental): In Arm E patients will receive treatment at the optimal energy and ALA dose determined form prior Arms.
  Interventions: Combination Product: SONALA-001(ALA) and MR-Guided Focused Ultrasound device (MRgFUS)

INTERVENTIONS:
Combination Product: SONALA-001(ALA) and MR-Guided Focused Ultrasound device (MRgFUS) — SONALA-001(ALA) given 5-7 hours prior to receiving the MRgFUS.
  Arms: Arm A Energy Dose-escalation; Arm B Time-escalation; Arm C ALA Dose-escalation; Arm E Optimal energy and ALA dose
Device: MR-Guided Focused Ultrasound device (MRgFUS) — MR-Guided Focused Ultrasound device (MRgFUS) alone
  Arms: Arm D MRgFUS alone

SUMMARY:
A Phase 0 single center, first in human, open-label study of ascending energy doses of sonodynamic therapy (SDT) utilizing the MRgFUS combined with intravenous ALA to assess safety and efficacy in up to 45 participants with recurrent HGG. Eligible participants who are scheduled for resection will be administered intravenous (IV) aminolevulinic acid HCl (ALA) approximately six to seven (6-7) hours prior to receiving sonodynamic therapy (SDT).

ELIGIBILITY:
Inclusion Criteria:

1. Arms A-D: Prior resection of histologically diagnosed high-grade gliomas (III and IV) defined as participants who have progressed on or following standard therapy as determined by the investigator. Arm E: Participant at first recurrence with an unmethylated HGG, has completed standard therapy and is not currently scheduled for resection.
2. Recurrence must be confirmed by diagnostic biopsy with local pathology review or contrast-enhanced MRI with positive perfusion.
3. Arms A-D (only): Have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with a volume of at least 6 cm3 and ≤ 20cm3 of targeted treatment area.
4. Age ≥18 at time of consent.
5. Have a performance status (PS) of ≤2 on the Eastern Cooperative Oncology (Group (ECOG) scale (Oken et al. 1982).
6. Has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility)

   Adequate bone marrow function:
   * absolute neutrophil count ≥1,000/mcL
   * Platelets (at time of surgery) ≥100,000/mcL
   * hemoglobin ≥8.0 g/dL Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator.

   Adequate hepatic and renal function:
   * total bilirubin ≤1.5 X ULN. Participants with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.
   * AST(SGOT) ≤3 X institutional ULN
   * ALT(SGPT) ≤3 X institutional ULN
   * GGT ≤3 X institutional ULN
   * Serum creatinine ≤1.5 X institutional ULN
7. Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant has had a hysterectomy.
8. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 3 months after the end of treatment administration.
9. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner and for an additional 1 month after the end of treatment administration. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner to prevent delivery of the drug via seminal fluid.
10. Participants who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to Day 1. A washout period of at least 14 days is required between last chemotherapy dose and Day 1 (provided the patient did not receive radiotherapy).
11. Participants who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and Day 1.
12. Ability to understand and the willingness to sign a written informed consent document (personally or by the legally authorized representative, if applicable).
13. Has voluntarily agreed to participate by giving written informed consent (personally or via legally authorized representative(s), and assent if applicable). Written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.
14. Willingness and ability to comply with scheduled visits, treatment plans, Lifestyle Considerations, laboratory tests and other procedures.

Exclusion Criteria:

1. Known active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
2. Have had a recent (≤3 months prior to first dose of study drug) transient ischemic attack or stroke.
3. Significant vascular disease (e.g. aortic aneurysm)
4. Evidence of bleeding diathesis or coagulopathy
5. Diagnosis of porphyria
6. Unstable angina and/or congestive heart failure within the last 6 months
7. Transmural myocardial infarction within the last 6 months
8. Serious and inadequately controlled cardiac arrhythmia
9. Acute exacerbation of chronic obstructive pulmonary disease
10. Inability to undergo MRI (e.g., presence of a pacemaker)
11. Pregnancy or breastfeeding
12. Has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study.
13. Simultaneous use of other potentially phototoxic substances (e.g. tetracyclines, sulfonamides, fluoroquinolones, hypericin extracts)
14. Hypersensitivity against porphyrins
15. Treatment with another investigational drug within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.
16. Has an Overall Skull Density Ratio of 0.45 (±0.05) or less as calculated from the screening CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Biological changes associated with the sonodynamic therapy | Intraoperatively 4, 7, or 14 days post sonodynamic therapy
  The percentage (%) of Cleaved Caspase-3 of the surgical tissue will be quantified and compared to intra-patient control specimens.
Radiographic evidence of tumor physiological imaging changes associated with SDT in recurrent HGG patients (Arm E) | Intraoperatively 4, 7, or 14 days post sonodynamic therapy
  Volume of enhancing tumor will quantified and compared between pre and post procedural scans (Arm E)

SECONDARY OUTCOMES:
Radiographic evidence of tumor physiological imaging changes associated with sonodynamic therapy | Pre and 14 Days Post-operative scan
  Dynamic Contrast Enhanced (DCE)-MRI data to quantify permeability
Radiographic evidence of tumor physiological imaging changes associated with sonodynamic therapy | Pre and 14 Days Post-operative scan
  Dynamic Susceptibility Contrast (DSC)-MRI data to quantify perfusion
Radiographic evidence of tumor physiological imaging changes associated with sonodynamic therapy | Pre and 14 Days Post-operative scan
  Diffusion Weighted Imaging (DWI) data to evaluate cellularity
To identify oxidative stress in tissue exposed to sonodynamic therapy in recurrent high-grade glioma patients. | Intraoperatively 2, 4, or 6 days post sonodynamic therapy
  To quantify markers for oxidative stress (Protein oxidation (Protein Carbonyl Content), Lipid peroxidation (4-hydroxynonenal and MDA), DNA damage (8-hydroxyguanosine),General (GSH, GSSG, Cys, CySS) in the brain tumor tissue (2-, 4- and 6-days post SDT) (both in SDT and control fractions)
Performance of MRgFUS | Day 1
  Percentage of SDT treatments in which the MRgFUS system works as planned
Performance of MRgFUS | Day 1
  Percentage of treatments in which procedure deviations were noted
Safety and Tolerability | up to 30 days after the last study dose
  Number and incidence of drug-related toxicity
Safety and Tolerability | up to 30 days after the last study dose
  Adverse device effects
To characterize the biological changes associated with sonodynamic therapy in recurrent high-grade glioma patients. | Intraoperatively 4, 7, or 14 days post sonodynamic therapy
  The percentage (%) of MIB-1 level, 4-hydroxynonenal (4-HNE) of the surgical tissue will be quantified and compared to intra-patient control specimens.
Overall Survival | 24 months
  Median overall survival
Progression-free survival | 6 months
  Number of patients who reach 6-month progression- free survival rate (PFS6)
Best Overall Response (BOR) | 24 months
  Proportion of patients with a BOR of CR or PR per RANO

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No